CLINICAL TRIAL: NCT04122599
Title: Melatonin for Prevention of Post Stroke Delirium
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 752/2018BO2
Record Dates: First submitted 2019-05-29; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2018-10

CONDITIONS: Post Stroke Delirium
Keywords: Melatonin
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Melatonin versus standard care (Other): Melatonin is tested versus standard care
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Melatonin for prevent post stroke delirium

SUMMARY:
Post stroke delirium is prevalent in 10-30% of all stroke patients. We aimed to investigate wether Melatonin 2mg may prevent post stroke delirium.

ELIGIBILITY:
Inclusion Criteria:

* all patients with stroke, TIA or ICH admitted to our stroke unit or intemdiate care unit
* Stroke / ICH /TIA onset <= 48h

Exclusion Criteria:

* RASS <=4
* severe dementia, psychosis or depression

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of delir prevalence | 3months

SECONDARY OUTCOMES:
Change of hospital stay | 3months
Change of antipsychotic drug administration | 3 months
Changed stay on stroke unit and/or intermediate care | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Neurologie, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No